CLINICAL TRIAL: NCT03780257
Title: A First-in-Human Study to Evaluate the Safety and Tolerability of QR-421a in Subjects With Retinitis Pigmentosa (RP) Due to Mutations in Exon 13 of the USH2A Gene
Brief Title: Study to Evaluate Safety and Tolerability of QR-421a in Subjects With RP Due to Mutations in Exon 13 of the USH2A Gene
Acronym: Stellar
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ProQR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PQ-421a-001; 2018-002433-38 (EudraCT Number)
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Retinitis Pigmentosa; Usher Syndrome Type 2; Deaf Blind; Retinal Disease; Eye Diseases; Eye Diseases, Hereditary; Eye Disorders Congenital; Vision Disorders
Keywords: Retinitis Pigmentosa; USH2A; RP; exon 13; RNA therapies; antisense oligonucleotide; exon skipping; STELLAR; IVT; mutations in exon 13 of the USH2A gene; NSRP
MeSH Terms: conditions — Retinitis Pigmentosa; Usher Syndromes; Retinal Diseases; Eye Diseases; Eye Diseases, Hereditary; Eye Abnormalities; Vision Disorders | interventions — Intravitreal Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QR-421a (Experimental): Single dose administration
  Interventions: Drug: QR-421a
- Sham-procedure (dose cohort 1&2 only) (Sham Comparator): Sham-procedure (no experimental drug administered)
  Interventions: Other: Sham-procedure (dose cohort 1&2 only)

INTERVENTIONS:
Drug: QR-421a — RNA antisense oligonucleotide for intravitreal injection
  Other Names: RNA antisense oligonucleotide for intravitreal injection
  Arms: QR-421a
Other: Sham-procedure (dose cohort 1&2 only) — Sham-procedure (no experimental drug administered)
  Other Names: Sham-procedure
  Arms: Sham-procedure (dose cohort 1&2 only)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of QR-421a administered via intravitreal injection (IVT) in subjects with Retinitis Pigmentosa (RP) due to mutations in exon 13 of the USH2A gene.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability of QR-421a administered via IVT in subjects with RP due to mutations in exon 13 of the USH2A gene. Subjects will receive one single IVT injection of QR-421a or sham-procedure in one eye (subject's worse eye) and will be followed up for 24 months.

Three dose levels of QR-421a will be evaluated: 50, 100, and 200 µg. Additional dose levels (eg, 25 or 400 µg) may be evaluated based on ongoing safety and efficacy data monitoring.

Initial dose cohorts will include subjects randomized to sham-procedure or treatment with QR-421a. Additional subjects may be allocated to treatment with QR-421a in subsequent or initial dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 years of age.
2. Clinical presentation consistent with RP with Usher syndrome type 2 or non-syndromic RP (NSRP), based on ophthalmic, audiologic, and vestibular examinations.
3. A molecular diagnosis of homozygosity or compound heterozygosity for 1 or more pathogenic exon 13 mutations in the USH2A gene, based on genetic analysis upon Sponsor approval.
4. Impairment of VF in the opinion of the Investigator, as determined by perimetry, with a continuous area of central field greater than or equal to 10 degrees diameter in any axis in the treatment eye, and evidence of functioning rods.
5. Willing and able to comply with the protocol, follow study instructions, attend study visits as required and complete all study assessments.
6. Willing and able to provide informed consent for participation prior to performing any study related procedures, and suitable verbal, auditory, written and/or tactile sign language communication as to allow informed consent to be obtained, in the opinion of the Investigator.
7. No limitations to SD-OCT image collection that would prevent high quality, reliable images from being obtained in both eyes as determined by the investigator.
8. Reliable perimetry measurements in both eyes, as described in the Imaging Manual and determined by the Investigator.
9. Clear ocular media and adequate pupillary dilation to permit good quality retinal imaging, as assessed by the Investigator.

Exclusion Criteria:

1. Presence of additional non-exon 13 USH2A pathogenic mutation(s) on the USH2A allele carrying the exon 13 mutation in subjects who are compound heterozygous for mutations in exon 13.
2. Presence of non-exon 13 USH2A pathogenic mutation(s) on both USH2A alleles in subjects who are homozygous for mutations in exon 13.
3. Presence of pathogenic mutations in genes (other than the USH2A gene) associated with Usher syndrome Type 2 or NSRP, or other inherited retinal degenerative diseases or syndromes.
4. Presence of any significant ocular or non-ocular disease/disorder (or medication and/or laboratory test abnormalities) which, in the opinion of the Investigator and with concurrence of the Medical Monitor, may either put the subject at risk because of participation in the study, may influence the results of the study, or the subject's ability to participate in the study. This includes but is not limited to a subject who: 1) is not an appropriate candidate for antisense oligonucleotide treatment, 2) has cystoid macular edema (CME) in the treatment eye. CME is permissible if stable for 3 months (with or without treatment). Past CME is permissible if resolved for more than 1 month.
5. History or presence of ocular herpetic diseases (including herpes simplex virus, varicella zoster or cytomegalovirus) in either eye.
6. Presence of any active ocular infection in either eye.
7. Presence of any of the following lens opacities in the treatment eye: cortical opacity ≥ +2, posterior subcapsular opacity ≥ +2, or a nuclear sclerosis ≥ +2, and which are: 1) clinically significant in the opinion of the Investigator, 2) would adequately prevent clinical and photographic evaluation of the retina.
8. History of amblyopia in the treatment eye.
9. Worse than 6 diopters myopia in the treatment eye.
10. Receipt within 3 months prior to Screening of any intraocular or periocular surgery (including refractive surgery), or an IVT injection or planned intraocular surgery or procedure during the course of the study.
11. Current treatment or treatment within the past 12 months with therapies known to influence the immune system (including but not limited to steroid implants, cytostatics, interferons, tumor necrosis factor (TNF)-binding proteins, drugs acting on immunophilins, or antibodies with known impact on the immune system). Subjects that have been treated with systemic steroids within the past 12 months or that require intermittent use of topical steroids may be considered for inclusion following approval by the Medical Monitor.
12. A history of glaucoma or an IOP greater than 24 mmHg in either eye that is not controlled with medication or surgery at the time of informed consent.
13. Use of any investigational drug or device within 90 days or 5 half-lives preceding the first dose of study medication, whichever is longer, or plans to participate in another study of an investigational drug or device during the PQ-421a-001 study period.
14. Any prior treatment with genetic or stem-cell therapy for ocular or non-ocular disease.
15. History of malignancy within 5 years prior to Screening, except adequately treated squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
16. Known hypersensitivity to antisense oligonucleotides or any constituents of the injection.
17. Pregnant and breastfeeding subjects. Females of childbearing potential and males must comply with using highly effective methods of contraception as defined in Section 6.2.2. Women of non-childbearing potential may be included without the use of adequate birth control, provided they meet the criteria in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of ocular adverse events (AEs) in the treatment and contralateral eye | 24 months
  Incidence and severity of ocular AEs
Incidence and severity of non-ocular AEs | 24 months
  Incidence and severity of non-ocular AEs

SECONDARY OUTCOMES:
Change in DAC perimetry | 24 months
  Change in Dark Adapted Chromatic (DAC) perimetry
Change in static perimetry | 24 months
  Change in static perimetry
Change in EZ area by SD-OCT | 24 months
  Change in Ellipsoid Zone (EZ) area/width by spectral domain optical coherence tomography (SD-OCT)
Change in BCVA | 24 months
  Change in Best Corrected Visual Acuity (BCVA)
Change in LLVA | 24 months
  Change in Low Luminance Visual Acuity (LLVA)
Change in microperimetry | 24 months
  Change in microperimetry
Changes in FST | 24 months
  Changes in Full-field Stimulus Threshold (FST)
Changes in FAF | 24 months
  Changes in Fundus autofluorescence (FAF)
AUC (0-∞) of QR-421a in serum | 24 months
  Area under the curve 0 hour to infinity [AUC(0-∞)] of QR-421a in serum
AUC (0-tlast) of QR-421a in serum | 24 months
  Area under the curve 0 hour to the final sample with a concentration greater than lower limit of quantification (LLOQ) [AUC(0-tlast)] of QR-421a in serum
Cmax of QR-421a in serum | 24 months
  Maximum concentration (Cmax) of QR-421a in serum
Tmax of QR-421a | 24 months
  Time to maximum concentration (Tmax) of QR-421a
T1/2 of QR-421a | 24 months
  Terminal elimination half-life (T1/2) of QR-421a
Serum clearance (CL) of QR-421a | 24 months
  Serum clearance (CL) of QR-421a
Volume of distribution (Vd) of QR-421a | 24 months
  Volume of distribution (Vd) of QR-421a

CONTACTS AND LOCATIONS:
Overall Officials: ProQR Medical Monitor, Study Director — ProQR Therapeutics; ProQR Clinical Trial Manager, Study Director — ProQR Therapeutics
Locations (7):
- United States (4):
  - Center for Clinical Research Operations, Massachusetts Eye and Ear, Boston, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Casey Eye Institute, Oregon Health & Science University, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
- Centre for Innovative Medicine, Department of Paediatric Surgery, Montreal Children's Hospital at the McGill University Health Centre, Montreal, Canada
- France (2):
  - Hôpital Gui de Chauliac - CHRU de Montpellier - Maladies Sensorielles Génétique, Montpellier
  - Centre de maladies rares CHNO des Quinze Vingts, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan CM, Tan TE, Jain K, Bylstra Y, Mathur RS, Tang RWC, Lee BJH, Jamuar SS, Kam S, Vithana EN, Lim WK, Fenner BJ. RETINITIS PIGMENTOSA ASSOCIATED WITH THE EYS C2139Y VARIANT : An Important Cause of Blindness in East Asian Populations. Retina. 2023 Oct 1;43(10):1788-1796. doi: 10.1097/IAE.0000000000003874. PMID 37418643
- [Derived] Miah KM, Hyde SC, Gill DR. Emerging gene therapies for cystic fibrosis. Expert Rev Respir Med. 2019 Aug;13(8):709-725. doi: 10.1080/17476348.2019.1634547. Epub 2019 Jun 27. PMID 31215818